CLINICAL TRIAL: NCT05708755
Title: Cytomegalovirus T Cell Immunity and Antiviral Prophylaxis Minimization in Lung Transplant Recipients
Brief Title: CMV Immunity Monitoring in Lung Transplant Recipients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Viracor Eurofins (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-01138
Record Dates: First submitted 2023-01-24; First posted 2023-02-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplant; Complications
MeSH Terms: interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Lung Transplant Recipients (Experimental): Lung transplant recipients with pre-transplant serological immunity to CMV. CMV-TCIP will be measured every 3 months post-transplant with antiviral prophylaxis discontinued when threshold is exceeded.
  Interventions: Device: Cytomegalovirus T Cell Immunity Panel (CMV-TCIP); Diagnostic Test: Donor-Derived Cell-Free DNA (dd-cfDNA) Assay; Drug: Valganciclovir

INTERVENTIONS:
Device: Cytomegalovirus T Cell Immunity Panel (CMV-TCIP) — Whole blood assay that evaluates T cell (CD4 and CD8) responses to cytomegalovirus (CMV) antigens via intracellular cytokine staining (ICS).
  Other Names: Viracor inSIGHT
Diagnostic Test: Donor-Derived Cell-Free DNA (dd-cfDNA) Assay — Determines the percentage of circulating cell-free DNA (cfDNA) in transplant recipients derived from donor grafts.
  Other Names: Viracor TRAC
Drug: Valganciclovir — Delivered as standard of care for post-lung transplant immunosuppression and infection prophylaxis. Started on the first day post-transplant at a standard dose of 900 mg daily and continued for 12 months. Dose adjustments may be necessary based on renal function and/or adverse effects (e.g. neutropenia). Dose adjustments are standard based on package insert recommendations.

SUMMARY:
The purpose of this study is to determine the safety and feasibility of using a laboratory test to guide duration of antiviral prophylaxis with valganciclovir (medication used to prevent viral infections) after lung transplant. The laboratory test, inSIGHT™ CMV T Cell Immunity Panel, measures patients' immune response to a common viral infection known as cytomegalovirus (CMV). The goal of this study will be to safely decrease how long patients need to take valganciclovir based on the results of the CMV T Cell Immunity Panel.

ELIGIBILITY:
Inclusion Criteria:

1. Received a lung transplant, or multi-organ transplant involving a lung at NYU Langone Health
2. Pre-existing serological immunity to CMV (R+)
3. Able and willing to provide informed consent

Exclusion Criteria:

1. Anti-thymocyte globulin induction immunosuppression
2. Perioperative desensitization
3. Pregnant or breastfeeding women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
CMV Viremia-Free Survival | Up to Month 12 Post-Transplant
  Defined as the the time from lung transplant until the first detection of CMV DNA in patients' blood.

SECONDARY OUTCOMES:
Incidence of CMV Viremia | Up to Month 12 Post-Transplant
  Number of times CMV DNA is detected in patients' blood.
Incidence of CMV Viremia Requiring Treatment | Up to Month 12 Post-Transplant
  Number of times treatment is necessary after CMV DNA is detected in patients' blood.
Incidence of Treatment-Resistant CMV Viremia | Up to Month 12 Post-Transplant
  Number of times treatment for CMV Viremia does not appear effective after CMV DNA is detected in patients' blood.
Incidence of Bacterial Pneumonia | Up to Month 12 Post-Transplant
  Measure of non-CMV post-transplant infectious complications.
Incidence of Aspergillus Infection | Up to Month 12 Post-Transplant
  Measure of non-CMV post-transplant infectious complications.
Incidence of Varicella Zoster Reactivation | Up to Month 12 Post-Transplant
  Measure of non-CMV post-transplant infectious complications.
Incidence of Neutropenia | Up to Month 12 Post-Transplant

CONTACTS AND LOCATIONS:
Overall Officials: Luis Angel, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No